CLINICAL TRIAL: NCT07036926
Title: Video-Based AI-Generated Peri-operative Instructions for Mitral Valve Surgery: A Randomized Controlled Trial on Health Outcomes and Patient Experience
Brief Title: Video-Based AI-Generated Peri-operative Instructions for Mitral Valve Surgery
Acronym: VIP-IMPACT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Joanna Chikwe (Other)
Collaborators: Cedars Sinai Medical Center, Los Angeles, USA (Unknown)
Responsible Party: Sponsor-Investigator, Joanna Chikwe, Professor & Chairman, Department of Cardiac Surgery, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00003876
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Mitral Valve Repair Surgery
Keywords: Artificial Intelligence; Video education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Peri-Operative Standard of Care and Artificial Intelligence Video Education Arm (Active Comparator): In this arm, patients will receive AI-generated, interactive, peri-operative video education program in addition to standard of care education
  Interventions: Other: Artificial Intelligence Video Education Arm
- Peri-Operative Standard of Care Education only Arm (No Intervention): In this arm, patients will receive the usual Standard of Care Peri-Operative Education

INTERVENTIONS:
Other: Artificial Intelligence Video Education Arm — A novel, AI-generated, interactive peri-operative video education program. AI videos will be personalized using medical record chart data, specifically the patient's name, surgery date, and past medical history.
  Arms: Peri-Operative Standard of Care and Artificial Intelligence Video Education Arm

SUMMARY:
1. The purpose of this study is to evaluate the impact of a novel, AI-generated, interactive peri-operative video education program on total unplanned healthcare utilization
2. The main procedures are questionnaires and watching a video.
3. The subject population includes patients who are scheduled for isolated mitral valve repair surgery.
4. All study procedures will occur here at Cedars Sinai.

DETAILED DESCRIPTION:
This study is a prospective, single center, randomized trial comparing an AI-generated peri-operative video education program to standard of care education (1:1 ratio) in patients undergoing MV repair. The trial will be conducted in Southern California. The primary aim of this study is to evaluate the impact of a novel, AI-generated, interactive peri-operative video education program on total unplanned healthcare utilization, defined as a composite of hospital readmissions, ED visits, and unplanned outpatient visits, among patients undergoing mitral valve (MV) repair compared with standard of care education. The secondary aim is to analyze the association between utilization of this educational program with hospital length of stay (LOS) and patient cardiovascular medication compliance compared to standard of care education. The tertiary aim of this trial is to evaluate a range of patient-centered outcomes (levels of anxiety, satisfaction, and discharge location) following receipt of this educational program compared with standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients ≥ 18 years planned for elective, isolated MV repair.
2. Provide Informed consent

Exclusion Criteria:

1. Insufficient computer/smart device knowledge. Children or caregivers can assist, but patients should be able to access their own email or text messages and navigate to the internet to use the provided AI generated educational intervention.
2. Inconsistent access to a smart device with internet connection throughout the study period.
3. Inability to speak, read, and understand English or Spanish
4. Need for any concomitant procedure at the time of MV repair

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Unplanned Healthcare Utilization events | From randomization to 30 days post-surgery
  includes the following events: unplanned (i.e. patient initiated) phone calls, emails, clinic visits, and ED visits.

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Chikwe, MD, Principal Investigator — Cedars-Sinai Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Steenbergen G, van Veghel D, van Lieshout D, Sperwer M, Ter Woorst J, Dekker L. Effects of Video-Based Patient Education and Consultation on Unplanned Health Care Utilization and Early Recovery After Coronary Artery Bypass Surgery (IMPROV-ED): Randomized Controlled Trial. J Med Internet Res. 2022 Aug 26;24(8):e37728. doi: 10.2196/37728. PMID 36018625
- [Background] Tromp F, Dulmen S, Weert J. Interdisciplinary preoperative patient education in cardiac surgery. J Adv Nurs. 2004 Jul;47(2):212-22. doi: 10.1111/j.1365-2648.2004.03081.x. PMID 15196195
- [Background] Kessels RP. Patients' memory for medical information. J R Soc Med. 2003 May;96(5):219-22. doi: 10.1177/014107680309600504. No abstract available. PMID 12724430
- [Background] Ljungqvist O, Francis NK, Urman RD, eds. Enhanced Recovery After Surgery: A Complete Guide to Optimizing Outcomes. Springer International Publishing; 2020. doi:10.1007/978-3-030-33443-7
- [Background] Grab M, Hundertmark F, Thierfelder N, Fairchild M, Mela P, Hagl C, Grefen L. New perspectives in patient education for cardiac surgery using 3D-printing and virtual reality. Front Cardiovasc Med. 2023 Mar 3;10:1092007. doi: 10.3389/fcvm.2023.1092007. eCollection 2023. PMID 36937915
- [Background] Watson DJ. Nurse coordinators and ERAS programs. Nurs Manage. 2018 Jan;49(1):42-49. doi: 10.1097/01.NUMA.0000527718.90264.89. No abstract available. PMID 29287049
- [Background] Brodersen F, Wagner J, Uzunoglu FG, Petersen-Ewert C. Impact of Preoperative Patient Education on Postoperative Recovery in Abdominal Surgery: A Systematic Review. World J Surg. 2023 Apr;47(4):937-947. doi: 10.1007/s00268-022-06884-4. Epub 2023 Jan 15. PMID 36641521
- [Background] Berkman ND, Sheridan SL, Donahue KE, Halpern DJ, Crotty K. Low health literacy and health outcomes: an updated systematic review. Ann Intern Med. 2011 Jul 19;155(2):97-107. doi: 10.7326/0003-4819-155-2-201107190-00005. PMID 21768583
- [Background] Fernandez-Castro M, Jimenez JM, Martin-Gil B, Munoz-Moreno MF, Martin-Santos AB, Del Rio-Garcia I, Redondo-Perez N, Lopez M. The influence of preoperative anxiety on postoperative pain in patients undergoing cardiac surgery. Sci Rep. 2022 Oct 1;12(1):16464. doi: 10.1038/s41598-022-20870-9. PMID 36183003
- [Background] Prado-Olivares J, Chover-Sierra E. Preoperatory Anxiety in Patients Undergoing Cardiac Surgery. Diseases. 2019 Jun 19;7(2):46. doi: 10.3390/diseases7020046. PMID 31248177
- [Background] Ramesh C, Nayak BS, Pai VB, Patil NT, George A, George LS, Devi ES. Effect of Preoperative Education on Postoperative Outcomes Among Patients Undergoing Cardiac Surgery: A Systematic Review and Meta-Analysis. J Perianesth Nurs. 2017 Dec;32(6):518-529.e2. doi: 10.1016/j.jopan.2016.11.011. Epub 2017 Apr 13. PMID 29157759